CLINICAL TRIAL: NCT03074669
Title: Internet-delivered Acceptance and Commitment Therapy for Reducing Anxiety Symptoms
Brief Title: Online Acceptance and Commitment Therapy for Reducing Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUTimisoara ACT-online
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Anxiety Disorder/Anxiety State
Keywords: Anxiety symptoms/disorders (OCD, PTSD, GAD, SAD, Panic)
MeSH Terms: conditions — Anxiety Disorders; Disease; Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT program (Experimental): Participants from the active treatment group will be granted access to seven modules that are structured like chapters of a self-help book adapted for the online environment. In addition, participants from the experimental arm will be guided by an on-line therapist throughout the program duration. The on-line therapists are graduate students in clinical psychology who work under the supervision of an experienced psychotherapist. Participants will be asked to fill in a series of self-report measures to monitor their anxiety and some ACT specific processes (i.e., acceptance, mindfulness, experiential avoidance) throughout the intervention.
  Interventions: Behavioral: ACT program
- Wait-list control group (No Intervention): During the first seven weeks, participants in the wait-list control group will only be asked to fill in a series of self-report measures to monitor their anxiety and some ACT specific processes (i.e., acceptance, mindfulness, experiential avoidance). Following the experimental group's completion of the program, participants in this group will also receive the intervention. All participants will be contacted 6 months after the intervention has concluded in order to conduct a follow-up assessment.

INTERVENTIONS:
Behavioral: ACT program — ACT program consists of seven modules that have been adapted for the online environment. Each module is structured like a therapy session with at least two homework assignments.
  Arms: ACT program

SUMMARY:
The main objective of this study is to test the effectiveness of an Internet-delivered Acceptance and Commitment Therapy (ACT) program in reducing anxiety symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness and level of acceptability of an Internet-delivered Acceptance and Commitment Therapy (ACT) program in reducing symptoms of anxiety. The effectiveness of the intervention will be compared with a wait-list control group using a randomized control trial (RCT) design. The participants with high / clinical levels of anxiety from the active treatment group will have the opportunity to read seven ACT modules and receive personalized feedback for their completed homework assignments.

The intervention will be delivered online and participants will have seven weeks to complete the seven modules (we might add one extra week of treatment for all participants in the event they need to compensate the treatment delays accumulated during the previous seven weeks).

ELIGIBILITY:
Inclusion Criteria:

* be fluent in Romanian
* be over 18 years of age
* have high levels of anxiety
* have access to an Internet-connected computer

Exclusion Criteria:

* suicidal ideation
* substance abuse
* severe psychiatric disorders
* a recent change in psychotropic medication (i.e., the dose has been changed within the last month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-05-15 (Estimated); Study Completion 2018-01-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Anxiety Sensitivity Index (ASI) | Change from Pre- to Post-Intervention (7 weeks), and Change from Post-intervention (week 7) to Follow-up (6 month post-intervention)
  The ASI was designed to identify fear of somatic and cognitive symptoms of anxiety due to a belief that these symptoms may be dangerous or harmful. The scale is unidimensional and the total score rages from 0 to 64. Low scores are associated with low levels of anxiety sensitivity, while high scores are associated with high levels of anxiety sensitivity.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The PSWQ was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score rages from 16 to 80. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.
Social Phobia Inventory (SPIN) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The SPIN was designed to measure participant's level of social phobia. The scale is unidimensional and the total score rages from 0 to 68. Low scores are associated with low levels of social phobia, while high scores are associated with high levels of social phobia.
Yale-Brown Obsessive Compulsive Scale (YBOCS) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The YBOCS was designed to measure participant's level of obsessions and compulsions (O&C). The scale total score rages from 0 to 40. Low scores are associated with low levels of O&C, while high scores are associated with high levels of O&C.
Panic Disorder Severity Scale - Self Report (PDSS-SR) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The PDSS-SR was designed to measure participant's level of panic. The scale is unidimensional and the total score rages from 0 to 28. Low scores are associated with low levels of panic, while high scores are associated with high levels of panic.
Post-Traumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual-5 (PCL-5) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The PCL-5 was designed to measure participant's level of post-traumatic stress. The scale is unidimensional and the total score rages from 0 to 80. Low scores are associated with low levels of post-traumatic stress, while high scores are associated with high levels of post-traumatic stress.
Beck Depression Inventory-II (BDI-II) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The BDI-II was designed to measure participant's level of depression. The scale is unidimensional and the total score rages from 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
Overall Anxiety Severity and Impairment Scale (OASIS) | Pre-intervention, week 2, week 4, week 6, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The OASIS was designed to measure participant's level of anxiety. The scale is unidimensional and the total score rages from 0 to 20. Low scores are associated with low levels of anxiety, while high scores are associated with high levels of anxiety.
Overall Depression Severity and Impairment Scale (ODSIS) | Pre-intervention, week 2, week 4, week 6, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)]
  The ODSIS was designed to measure participant's level of depression. The scale is unidimensional and the total score rages from 0 to 20. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression
Acceptance and Action Questionnaire 2 (AAQ2) | Pre-intervention, week 2, week 4, week 6, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The AAQ2 was designed to measure of ACT's model of mental health and behavioral effectiveness. Scores range from 7 to 49 points, with high scores indicating greater experiential avoidance and immobility.
Mindful Attention Awareness Scale (MAAS) | Pre-intervention, week 2, week 4, week 6, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness. Higher scores reflect higher levels of dispositional mindfulness.
Believability of Anxious Feelings and Thoughts Questionnaire (BAFT) | Pre-intervention, week 2, week 4, week 6, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The BAFT is a 16 item measure of cognitive fusion with anxious thoughts and feelings. Scores range from 16 to 112.
Brief Multidimensional Experiential Avoidance Questionnaire (BMEAQ) | Pre-intervention, week 2, week 4, week 6, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The 15 item BMEAQ was developed to measure the tendency to avoid negative internal experiences .
Quality of Life Inventory (QOLI) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The QOLI assesses an individual's quality of life through self-report of the importance they attach to each of 16 life domains. Each item is rated twice according to a) the importance to the overall happiness and satisfaction (0 = not at all important, 1 = important, 2 = extremely important) and b) satisfaction with the area ( -3 = very dissatisfied to +3 = very satisfied). The QOLI is a unidimensional scale with a continuous score that rages from -6 to +6, with negative score indicating a low life quality and the positive score indicating a high life quality.
Work and Social Adjustment Scale (WSAS) | Pre-intervention, Post-Intervention (7 weeks) and at Follow-up (6 month post-intervention)
  The WSAS measures impaired functioning.The maximum score of the WSAS is 40 with lower scores suggesting better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Tudor Tulbure, PhD, Principal Investigator — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No
Data will be process only at the group level. No individual data will be shared to third parties.